CLINICAL TRIAL: NCT01469806
Title: Zimmer(R) Gender Solutions(TM) Patello-Femoral Joint Prothesis Used Within the Knee Registry Protocol
Brief Title: Patello-Femoral Joint Post Market Clinical Follow-up Within the Knee Registry
Acronym: PFJPMCF
Status: Withdrawn | Type: Observational
Why Stopped: Suspended pending internal review/direction of the company's focus. No sites ever engaged or collected data.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 04-400; 90-112 (Other: Zimmer, Inc)
Record Dates: First submitted 2011-10-24; First posted 2011-11-10 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2012-03

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 - PFJ: Patients who require primary partial knee arthroplasty of the patello-femoral joint.
  Interventions: Device: Zimmer Gender Solutions PFJ Knee Prosthesis

INTERVENTIONS:
Device: Zimmer Gender Solutions PFJ Knee Prosthesis — Partial knee arthroplasty of the patello-femoral joint

SUMMARY:
The primary objective of the Registry is to allow for tracking of FDA approved and/or cleared knees used in primary, revision, unicompartmental or partial total knee arthroplasty (TKA). Second, it is our desire to assist orthopaedic surgeons in obtaining and evaluating radiographic and functional outcomes data on their PFJ patients using current published guidelines. Third, within this Registry, subsets of data on newer technology are being collected for the purpose of future publications. The Patello-Femoral Joint Post Market Clinical (PFJ PMCF) study is one such subset.

DETAILED DESCRIPTION:
To obtain preoperative, operative and postoperative clinical outcomes data for the Zimmer Gender Solutions PFJ Knee Prosthesis used in primary partial knee arthroplasty such as knee scoring and patient satisfaction such collection using Patient Questionaire and SF-12 forms. Kaplan-Meir survivorship analysis of the device will be performed. Radiographic analysis of the device will also be performed at 1, 2, 3, 5, 7, and 10 year follow-up. It is planned that the resultant data will be pooled and published by the evaluating surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than 18 years of age;
* Patient selection is without bias to race or gender;
* Patient is in stable health and able to undergo surgery;
* Patient has patellofemoral joint(s) affected by disease process and/or injury and qualifying for primary unilateral or bilateral replacement of the femoral trochlea based a primary diagnosis of at least one of the following:

  * Osteoarthritis
  * Traumatic Arthritis
  * Polyarthritis
  * Severe Chondrocalcinosis
  * Salvage of previously failed surgical attempts (e.g., arthroscopy, lateral release, cartilage transplantation)
  * History of patellar dislocation or patella fracture
  * Dysplasia-induced patellofemoral degeneration
* Patient is willing and able to cooperate in prescribed post-operative therapy;
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent;
* Patient has participated in the Informed Consent process and has signed an IRB approved Informed Consent.
* Patient has not history of previous prosthetic replacement device(s) of any type in the affected knee joint;
* Independent of study participation, patient is scheduled to receive treatment using a Zimmer Gender Solutions Patellofemoral Joint Prosthesis (PFJ).

Exclusion Criteria:

* Patient with an acute, chronic, local or systemic infection;
* Patient is skeletally immature;
* Patient is pregnant;
* Patient is a prisoner, mentally incompetent or anticipated to be non-compliant. Patient has a known allergy to one of the constituents of the implant, e.g. cobalt, chromium, nickel, etc.;
* Patient has Rheumatoid Arthritis (RA) AND an ulcer of the skin OR a history of recurrent breakdown of the skin;
* Patient has neuropathic arthropathy, neuromuscular disorder, neurologic condition, vascular disorder, systemic disease and/or other condition that affects lower limb function and/or could contribute to prosthesis instability, prosthesis fixation failure, and/or complications in postoperative care;
* Patient has a Body Mass Index (BMI) greater than 40;
* Patient has insufficient native bone stock in the operative joint (e.g. osteoporosis, osteonecrosis, tumors, cysts, etc.). Note: Bone void fillers are NOT considered native bone stock, even if autograft is used;
* Patient has severe instability, maltracking, or malalignment of the patella, patellofemoral, and/or tibiofemoral joints;
* Patient has patellectomy of the affected joint, including previous patellectomy, patellectomy performed simultaneous to study PFA, or scheduled patellectomy;
* Patient has insufficient menisci and/or ligament structures (e.g. non-functional/absent ACL and/or PCL);
* Patient exhibits tibiofemoral degeneration and/or Outerbridge grade greater than or equal to 3 in EITHER:

  * one (medial or lateral) tibiofemoral compartment that is not treated with a simultaneous compatible Zimmer unicompartmental knee replacement; OR
  * both (medial AND lateral) tibiofemoral compartments, regardless of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient has patellofemoral joint(s) affected by disease process and /or injury and qualifying for primary unilateral or bilateral replacement of the femoral trochlea based a primary diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Long-term Device survivorship for publication | 10 Years

SECONDARY OUTCOMES:
Radiographic analysis of enrolled subjects | 10 years

IPD SHARING:
Plan to Share IPD: No